CLINICAL TRIAL: NCT02718157
Title: Prospective Study for Clinical Validation of the Molecular-Based GenePOC GBS Assay for the Detection of the Cfb Gene From Streptococcus Agalactiae Strains in Vaginal/Rectal Swab Specimens, After Lim Broth Enrichment, From Pregnant Women
Brief Title: Validation of the GenePOC GBS Assay for the Detection of the Cfb Gene From Streptococcus Agalactiae Strains
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meridian Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GenePOC-GBS_clinical-01
Record Dates: First submitted 2016-03-15; First posted 2016-03-24 (Estimated); Results first posted 2018-12-13 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2018-11

CONDITIONS: Streptococcus Agalactiae Infection
Keywords: Polymerase Chain Reaction (PCR); GBS; Streptococcus agalactiae; Antepartum women
MeSH Terms: conditions — Streptococcal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes

ARMS (1):
- Accuracy Testing (Experimental): Comparison between GenePOC PCR and Reference Method
  Interventions: Device: Comparison between GenePOC PCR and Reference Method

INTERVENTIONS:
Device: Comparison between GenePOC PCR and Reference Method — Antepartum women swab specimen incubated in Lim Broth will be tested with the GenePOC GBS test on the GenePOC Instrument. The results will be compared to Reference Method defined as incubated Lim broth subcultured onto blood agar plate for observation of a Streptococcus agalactiae strain.

SUMMARY:
The primary purpose of this clinical investigation is to verify the performance of the GenePOC GBS Assay on the GenePOC Instrument. This will be achieved by comparing the Assay to the a Culture, a conventional method for detection of Streptococcus agalactiae in vaginal/rectal swab specimens from antepartum women.

DETAILED DESCRIPTION:
The GenePOC GBS Test performed on the GenePOC System is a qualitative in vitro diagnostic (IVD) test designed to detect Group B Streptococcus (GBS) DNA from vaginal/rectal swabs from antepartum women following enrichment in Lim broth for 18-24 hours.

The GenePOC GBS Test utilizes automated sample preparation and real-time polymerase chain reaction (PCR) to detect a cfb gene sequence specific to the Streptococcus agalactiae genome. The GenePOC GBS Test is indicated for the identification of antepartum GBS colonization and does not provide susceptibility results. Culture isolates are needed for performing susceptibility testing as recommended for penicillin-allergic women.

The GenePOC GBS is an IVD system is comprised of the GenePOC Diagnostics System and the GenePOC Group B Step [GBS] Test, the components of which are:

1. Instrument
2. GBS disposable microfluidic cartridges (PIE) (described in this document as PIEs because of the shape of the cartridge)
3. GBS Sample Buffer Tube (SBT)
4. Sample Transfer Device (STD).

The GenePOC Instrument is fully automated and integrates sample lysis, dilution, amplification and detection of the target sequence in complex samples using real-time Polymerase chain reaction (rtPCR). User intervention is only required for discharging the patient sample into the SBT (sample Buffer Tube), transferring the sample into the PIE and for loading/unloading the PIEs into the instrument. The GenePOC instrument consists of a rotor to spin the PIEs, temperature control, fluorescence detection, a tactile user-friendly interface, two barcode readers, and integrated firmware and software to deliver results to the user. The PIE is a closed system that prevents the risk of contamination.

Lim Broth is used for the selective enrichment of group B streptococci (Streptococcus agalactiae). An aliquot of the broth is mixed with GenePOC Sample Buffer Tube Reagent (SBT), after which a sample is transferred to the GenePOC GBS PIE. The GenePOC GBS PIE is then automatically processed by the GenePOC Instrument.

On completion of a run, the user removes the processed PIEs from the instrument and discards them according to local biological waste management procedures.

One GenePOC instrument per site will be allocated. The purpose of the clinical investigation is to enroll sufficient specimens from four (4) Clinical Centers to obtain a total of 150 specimens positive for GBS based on the Reference Method final result.

Subject Informed consent is not required for this clinical trial as the testing will be performed on excess de-identified specimens only.

ELIGIBILITY:
Inclusion Criteria:

* Antepartum pregnant women
* 18 years old and more
* Being at a gestation period of 35 to 37 weeks.
* Vaginal/rectal swab specimen
* Transport and storage times, and conditions (e.g. room temperature and/or refrigerated) within the labeled indications.

  * Fresh specimens available to be tested with the GenePOC GBS System within 96 hours (4 days) of collection if kept at 2-25°C
  * Fresh specimens must be tested with the Reference Method within 96 hours (4 days) of collection if kept at 2-25°C
* The GenePOC GBS System and the Reference Method will be performed according to the GenePOC GBS Investigation Documents.
* Materials use within their expiration date

Exclusion Criteria:

* Non pregnant women
* Less than 18 years old
* Gestation not between 35-37 weeks
* Transport and storage times and conditions that exceed these Study Protocol requirements
* The GenePOC GBS System and the Reference Method not performed according to the GenePOC GBS Investigation Documents
* Materials used beyond their expiration date
* Specimens without all test results required by this Study Protocol. Specimens that are inadvertently entered into the study that do not meet the specimen inclusion criteria will be made non-compliant.
* The GenePOC GBS System and the Reference Method not performed according to the GenePOC GBS Investigation Documents.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 771 (Actual)
Dates: Start 2016-08-10 (Actual); Primary Completion 2017-02-07 (Actual); Study Completion 2017-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrice Allibert, Study Director — Meridian Bioscience, Inc.
Locations (4):
- United States (2):
  - Detroit Medical Center University Laboratories, Detroit, Michigan
  - Tricore Laboratory University of New Mexico, Albuquerque, New Mexico
- Canada (2):
  - Mount Sinai Hospital Joseph and Wolf Lebovic Health Complex, Toronto, Ontario
  - CHU de Québec - Université Laval, Québec

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Accuracy Testing
Started | 771
Completed | 609
Not Completed | 162

BASELINE CHARACTERISTICS:
Arm/Group | Accuracy Testing
Number analyzed (Participants) | 771
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 771
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 771
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 238
  United States | 533

OUTCOME MEASURES:

1. Primary Outcome: Performance Characteristics
Description: To establish the performance characteristics of the GenePOC GBS System for its use in determining the presence of GBS in vaginal/rectal swab, after Lim Broth enrichment, specimens from antepartum pregnant women. Sensitivity and specificity will be established in comparison to the Reference Method.
  Sensitivity performance results from the comparison of specimens being reported as positive by both method against the total number of specimen reported as positive on the Reference Method only. Sensitivity is reported as a percentage (i.e. concondant positives / concordant positive + discordant positive ([False Negative]).
  Specificity performance results from the comparison of specimens being reported as negative by both method against the total number of specimen reported as negative on the Reference Method only. Specificity is reported as a percentage (i.e. concondant negatives / concordant negatives + discordant negatives ([False Positive]).
Time Frame: At the time of the results with Reference Method is confirmed, up to 6 months
Measure: Number (95% Confidence Interval); unit: percentage of specimens
Arm/Group | Accuracy Testing
Number analyzed (Participants) | 771
percentage of specimens
  Sensitivity | 95.9 [91.7 to 98.0]
  Specificity | 95.5 [93.5 to 96.9]

2. Secondary Outcome: Positive and Negative Predictive Values
Description: To estimate the Positive and Negative Predictive Values (PPV and NPV) of the GenePOC GBS System.
  PPV results from the comparison of specimens being reported as positive by both method against the total number of specimen reported as positive on the Investigational test only. PPV is reported as a percentage (i.e. concondant positives / concordant positive + discordant positive ([False Positive]).
  NPV results from the comparison of specimens being reported as negative by both method against the total number of specimen reported as negative on the Investigational test only. NPV is reported as a percentage (i.e. concondant negatives / concordant negatives + discordant negatives ([False Negative]).
Time Frame: At the time of the results with Reference Method is confirmed, up to 6 months
Measure: Number (95% Confidence Interval); unit: percentage of specimens
Arm/Group | Accuracy Testing
Number analyzed (Participants) | 771
percentage of specimens
  PPV | 85.8 [80.1 to 90.0]
  NPV | 98.8 [97.5 to 99.4]

3. Secondary Outcome: Unresolved Sample Results
Description: To estimate the rate of unresolved results for the GenePOC GBS System due to Sample Processing control failure (unresolved sample results).
Time Frame: At the time of the results with Reference Method is confirmed, up to 6 months
Measure: Number (95% Confidence Interval); unit: percentage of Unresolved
Arm/Group | Accuracy Testing
Number analyzed (Participants) | 771
percentage of Unresolved | 0.74 [0.34 to 1.60]

4. Secondary Outcome: Indeterminate Sample Results
Description: To estimate the rate of indeterminate results for the GenePOC GBS Test due to an Instrument failure (indeterminate sample results).
Time Frame: At the time of the results with Reference Method is confirmed, up to 6 months
Measure: Number (95% Confidence Interval); unit: percentage of Indeterminates
Arm/Group | Accuracy Testing
Number analyzed (Participants) | 771
percentage of Indeterminates | 1.48 [0.85 to 2.57]

ADVERSE EVENTS:
Time Frame: From 26 August 2016 to 01 November 2016. Adverse event were assessed at the time of individual patient enrollment and participation, which lasts approximately 1-2 minutes at most.
Description: Adverse event procedures were established at each site, but no adverse event was observed nor reported during the enrollment period.
Arm/Group | Accuracy Testing
All-Cause Mortality (participants affected / at risk) | 0/771
Serious Adverse Events (participants affected / at risk) | 0/771
Other Adverse Events (participants affected / at risk) | 0/771

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-05): https://cdn.clinicaltrials.gov/large-docs/57/NCT02718157/Prot_SAP_000.pdf